CLINICAL TRIAL: NCT04229979
Title: A Randomized, Open-Label Study of the Efficacy and Safety of Galinpepimut-S (GPS) Maintenance Monotherapy Compared to Investigator's Choice of Best Available Therapy in Subjects With Acute Myeloid Leukemia Who Have Achieved Complete Remission After Second-Line Salvage Therapy
Brief Title: Galinpepimut-S Versus Investigator's Choice of Best Available Therapy for Maintenance in AML CR2/CRp2
Acronym: REGAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sellas Life Sciences Group (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLSG18-301
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: maintenance; complete remission; overall survival; galinpepimut-S; randomized; Wilms Tumor-1 protein
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Pathologic Complete Response | interventions — Azacitidine; venetoclax; Decitabine; Cytarabine; Observation; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Monatide (IMS 3015)

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, randomized, parallel group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galinpepimut-S + Montanide + GM-CSF (Experimental): Galinpepimut-S injections will be administered as follows, until disease relapse:
  1. First 6 galinpepimut-S injections: every 2 weeks (Weeks 0 - 10) followed by a 4-week period of no treatment. The first series of 6 injections of galinpepimut-S define the initial immunization induction phase.
  2. Injections 7 to 12: every 4 weeks (Weeks 14 - 34) followed by a 6-week period of no treatment. The second series of injections of galinpepimut-S define the early immune booster phase.
  3. Injections 13 to 15: every 6 weeks (Weeks 40 - 52). The third series of injections of galinpepimut-S define the late immune booster phase.
  4. Injections 16-20: every 2 months (in Year 2).
  5. Injection 21 and thereafter: every 3 months (in Year 3). Y2 and Y3 define the maintenance phase.
  Note: Galinpepimut-S is admixed with Montanide adjuvant before administered as a subcutaneous injection. GM-CSF is administered two days before and on the same day as the galinpepimut-S + Montanide injection.
  Interventions: Biological: Galinpepimut-S; Biological: GM-CSF; Other: Montanide
- Best Available Therapy (Active Comparator): Four options, as monotherapy or as combination of agents listed below, (per treating investigator's choice):
  1. Observation (whereby palliative management with hydroxyurea is allowed), or
  2. HMA (decitabine or azacitidine), and/or
  3. Venetoclax, and/or
  4. Low-dose ara-C
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Decitabine; Drug: Cytarabine; Other: Observation

INTERVENTIONS:
Biological: Galinpepimut-S — Galinpepimut-S admixed with the adjuvant Montanide following specified schedule
  Other Names: SLS-001; GPS
  Arms: Galinpepimut-S + Montanide + GM-CSF
Drug: Azacitidine — injection
  Arms: Best Available Therapy
Drug: Venetoclax — tablet
  Arms: Best Available Therapy
Drug: Decitabine — injection
  Arms: Best Available Therapy
Drug: Cytarabine — injection
  Other Names: Ara-C
  Arms: Best Available Therapy
Other: Observation — palliative management
  Arms: Best Available Therapy
Biological: GM-CSF — subcutaneous injection
  Other Names: sargramostim
  Arms: Galinpepimut-S + Montanide + GM-CSF
Other: Montanide — adjuvant
  Arms: Galinpepimut-S + Montanide + GM-CSF

SUMMARY:
To assess the safety and efficacy of galinpepimut-S (GPS) compared with investigator's choice of best available therapy (BAT) on overall survival (OS) in subjects with acute myeloid leukemia (AML) who are in second or later complete remission (CR2) or second or later complete remission with incomplete platelet recovery (CRp2).

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized, parallel groups study of galinpepimut-S (GPS) vs. best available treatment (BAT) in patients with AML in second complete remission (CR2) or in second complete remission with incomplete platelet recovery (CRp2). All patients will have their historical bone marrow samples and/or peripheral blood drawn during screening stained for WT1 via IHC and/or analyzed via PCR by central pathology review. The primary goal of the study will be to demonstrate an advantage for GPS in overall survival in these patient populations. The study will enroll approximately 140 patients and will be conducted at about 110 investigational sites. Patients will be randomized 1:1 to GPS or BAT stratified by whether they are in CR2 or CRp2, their cytogenetic risk at diagnosis (poor vs all other), whether they harbor minimal residual disease (MRD), and the duration of CR1 of less than one year or one year or more.

Patients on the BAT arm may be treated with 1. observation (whereby palliative management with hydroxyurea is allowed), 2. a hypomethylating agent (decitabine or azacitidine), 3. venetoclax and/or 4. low-dose ara-C. Patients whose remission in CR2 can be maintained with molecularly targeted agents (e.g. FLT-3 or IDH inhibitors) per investigator's determination will not be eligible. However, there are no restrictions on prior use of any agents in the CR1 setting. Patients cannot receive GPS as an adjunct therapy to any other agents.

Patients on the GPS arm will receive 70 μg of sargramostim (GM-CSF) on Day -2 and Day 1 before each injection of GPS. The first two administrations of GM-CSF will take place at the same anatomical site as the planned administration of GPS within each treatment cycle. GPS will be administered as an immunization induction every 2 weeks for 6 administrations (Weeks 0 - 10); this will be followed by a 4-week period of no treatment. Treatment will then resume for 6 administrations as an initial booster phase every 4 weeks (Weeks 14 - 34) which will again be followed by a period of no treatment lasting 6 weeks. GPS will be resumed after this period as a second booster phase and will be administered every 6 weeks (Weeks 40 - 52). Patients who remain in remission after 52 weeks will receive treatment every 2 months (Q2M) in the second year of treatment. Patients who remain in remission after 2 years will be treated every 3 months (Q3M) until disease relapse. Following each administration of GM-CSF or GPS, patients will be observed for approximately 30 minutes. An End of Treatment visit will be conducted 30 days following the last dose of GPS. Patients will then enter the long-term follow-up portion of the trial where they will be followed for recurrence of leukemia and overall survival.

To ensure a comparable level of observation, patients randomized to the BAT arm will be seen every 4 weeks through Week 52.

All patients will undergo bone marrow aspirates and biopsies at screening, Week 12, Week 52, and end of treatment or relapse. Bone marrow examinations will then be repeated as clinically indicated. Patients will be assessed for safety at each clinic encounter. The primary endpoint will be overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and provide signed informed consent for the study that fulfills Institution Review Board (IRB) guidelines.
2. Male or female patients ≥18 years of age on the day of signing informed consent.
3. Must have a diagnosis of AML according to the WHO criteria (primary/de novo or secondary, including treatment-related [e.g., due to prior anthracycline use], as well as cases due to progression of antecedent hematological disorder [e.g., MDS, MPN, or MDS/MPN 'overlap' syndrome).
4. Must be in second morphological complete remission (with or without platelet recovery; CR2/CRp2) for relapsed AML based upon the CRp criteria as follows:

   1. <5% myeloblasts in bone marrow
   2. Absence of Auer rods
   3. Absence of circulating peripheral blasts
   4. Peripheral blood absolute neutrophil count (ANC) >1000 cells/µL
   5. Peripheral blood platelet count >20,000/µL
   6. Absence of extramedullary disease
5. Patients must have > 300 lymphocytes/ μL.
6. Must not be candidates at the time of study entry for allogeneic stem cell transplant (Allo-SCT) due to intercurrent medical conditions, patient's preference or lack of an available donor.
7. Must have received the last dose of re-induction antileukemic therapy at least 4 weeks or ten half-lives of induction therapy (whichever is shorter) prior to receiving study treatment.
8. Must be consented within 6 months of having achieved CR2/CRp2 or later.
9. Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2 or 3.
10. Must have an estimated life expectancy >6 months.
11. If female, is postmenopausal (at least 12 sequential months of amenorrhea) or surgically sterile. Females of childbearing potential must have a negative pregnancy test
12. Female patients of childbearing potential who are heterosexually active and male patients with female sexual partners of childbearing potential must agree to use an effective method of contraception (e.g., oral contraceptives, double-barrier methods such as a condom and a diaphragm, intrauterine device) during the study and for 4 to 6 months (depending on treatment) following the last dose of study medication, or to abstain from sexual intercourse for this time; a woman not of childbearing potential is one who has undergone bilateral oophorectomies or who is post- menopausal, defined as the absence of menstrual periods for 12 consecutive months.
13. Must have recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5 Grade 0 or 1 after completion of prior AML therapy with the exception of the platelet count requirements (i.e., as long as peripheral blood platelet count is >20,000/µL).
14. Must not have end stage renal disease.
15. Must have adequate hepatic function defined as a serum total bilirubin <2 × ULN (except for Gilbert's syndrome, which will allow bilirubin ≤3.0 mg/dL), and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN.
16. Must be willing and able to return to the clinical site for adequate follow-up and to comply with the protocol as required.

Exclusion Criteria:

1. For subjects randomized to GPS maintenance monotherapy:

   1. Continuation of any agents administered as part of induction of CR2/CRp2 or later
   2. Receiving any concurrent anti-AML systemic therapy
   3. Prior clinically significant allergic reaction to Montanide, sargramostim (GM-CSF) or filgrastim (granulocyte colony stimulating factor [G-CSF]).
   4. Received any consolidation and/or maintenance antileukemic therapy, investigational agent, systemic corticosteroid therapy, or other immunosuppressive therapy within 4 weeks prior or 10 half lives, whichever is shorter prior to receiving study treatment. Systemic corticosteroids for chronic conditions (at doses ≤10 mg/day of prednisone or equivalent) or permitted, as are inhalational, intra-ocular, intra-articular and topical corticosteroids as well as any corticosteroids or other immunosuppressive therapies that do not act systemically (e.g. budesonide) at any dose level.
2. Imminently planned hematopoietic stem cell transplant (autologous or allogeneic, with any degree of match donor).
3. Acute promyelocytic leukemia or any morphologic and molecular variants, inclusive.
4. Serious concurrent illness that in the opinion of the Investigator would pose an undue risk to the subject being participating in the clinical study.
5. Currently have, central nervous system leukemia.
6. Received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Vaccines for Covid-19 used under an EUA, are considered an authorized (though not an approved or cleared) medical product for use in clinical care. Vaccines used for the prevention of Covid-19 are allowed to be used.
7. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks, or in the case of drugs 10 half lives, whichever is shorter, prior to the first dose of study treatment.
8. Patients who had an SCT after their most recent re-induction that resulted in CR2 or CRp2 or later are not eligible. Patients with prior SCT are allowed only if they had SCT prior to their latest re-induction or achieved CR by means of transplant ("hot transplant").
9. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy exceeding 10 mg daily of prednisone equivalent within 7 days prior the first dose of study drug. The use of physiologic doses of corticosteroids and/or immunosuppressive agents may be approved after consultation with the Sponsor. Steroids taken as short-term therapy (≤ 7 days) for antiemesis are permissible.
10. Known additional malignancy that is progressing or has required active treatment within the past 5 years, even if currently inactive or unapparent.
11. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
12. Known hypersensitivity to Montanide or vaccine adjuvants.
13. Previous clinically significant systemic allergic reaction to Montanide, sargramostim (GM-CSF), or filgrastim (G-CSF).
14. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
15. Active life threatening infection requiring systemic therapy.
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. This includes any serious, intercurrent, chronic, or acute illness, such as cardiac disease (New York Heart Association [NYHA] class III or IV), hepatic disease, or other illness considered by the investigator as an unwarranted high risk for investigational drug treatment.
17. Known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
18. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 4 to 6 months (depending on treatment) after the last dose of study treatment.
19. Has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
OS | 5 years
  Interval between randomization and death from any cause

SECONDARY OUTCOMES:
LFS | 5 years
  Interval between randomization and recurrence of leukemia or death from any cause
OS rate (%) | At 6, 9 and 12 months
  Percentage of patients surviving
LFS rate (%) | At 6, 9, and 12 months
  Percentage of patients surviving and being free of leukemic relapse

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Cicic Chief Development Officer, MD, Study Director — Sellas Life Sciences Group
Locations (73):
- United States (17):
  - O'Neal Comprehensive Cancer Center, Birmingham, Alabama
  - UCLA Medical Hematology and Oncology, Los Angeles, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Colorado Blood Cancer Institute - SCRI - PPDS, Denver, Colorado
  - Mayo Clinic Jacksonville Florida, Jacksonville, Florida
  - Augusta University, Augusta, Georgia
  - Rush University Cancer Center, Chicago, Illinois
  - Tulane Cancer Center - Liberty, New Orleans, Louisiana
  - Northwell Health Cancer Institute, Lake Success, New York
  - New York Medical College, Valhalla, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Bon Secours St. Francis Cancer Center, Greenville, South Carolina
  - Baylor Scott and White Research Institute, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Gainesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- France (9):
  - CHU Amiens-Picardie - Hopital Sud, Amiens
  - CHU Angers, Angers
  - CHU de Caen, Caen
  - CHU de Grenoble, Grenoble
  - Hôtel Dieu - Nantes, Nantes
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Leipzig, Leipzig
  - Universitätsklinik Rostock, Rostock
- Greece (10):
  - University General Hospital of Alexandroupoli, Alexandroupoli
  - General Hospital of Athens "Evaggelismos", Athens
  - General Hospital of Athens "Laiko", Athens
  - General Hospital of Athens "G. Gennimatas", Athens
  - General Hospital of Athens "Ηippokration", Athens
  - University General Hospital "Attikon", Chaïdári
  - General Hospital of Thessaloniki "G. Papanikolaou", Chortiatis
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Patras, Rio
  - University General Hospital of Thessaloniki "Ahepa", Thessaloniki
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Petz Aladár Egyetemi Oktató Kórház, Győr
  - Pécsi Tudományegyetem, Pécs
- India (5):
  - Malabar Cancer Centre, Kannur, Kerala
  - Yashoda Hospital, Hyderabad
  - Fortis Hospital, Ludhiāna
  - All India Institute of Medical Sciences, New Delhi
  - State Cancer Institute, Indira Gandhi Institute of Medical Sciences, Patna
- Poland (10):
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne Klinika Hematologii i Transplantologii, Gdansk
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Swietokrzyskie Centrum Onkologii, Kielce
  - Wojewodzki Szpital Specjalistyczny w Legnicy, Legnica
  - Zaklad Opieki Zdrowotnej MSW z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - Szpital Wojewodzki w Opolu, Opole
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Słomniki
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Serbia (2):
  - University Clinical Center of Serbia, Belgrade
  - Clinical Centre of Vojvodina, Novi Sad
- Spain (9):
  - Hospital de San Pedro de Alcantara, Cáceres
  - C.H. Regional Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Clinica Universidad Navarra, Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (5):
  - Changhua Christian Hospital, Chang-hua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jamy O, Cicic D. REGAL: galinpepimut-S vs. best available therapy as maintenance therapy for acute myeloid leukemia in second remission. Future Oncol. 2025 Jan;21(1):73-81. doi: 10.1080/14796694.2024.2433935. Epub 2024 Nov 28. PMID 39606837